CLINICAL TRIAL: NCT01241383
Title: Effect of Bosentan in the Course of Scleroderma Renal Crisis
Brief Title: Effect of Bosentan in Scleroderma Renal Crisis
Acronym: ScS-REINBO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P081217
Record Dates: First submitted 2010-11-12; First posted 2010-11-16 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2015-10

CONDITIONS: Scleroderma Renal Crisis
Keywords: Scleroderma renal crisis; angiotensin converting enzyme inhibitors; bosentan; endothelin receptor antagonist
MeSH Terms: interventions — Bosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bosentan (Experimental): Bosentan 62.5mg bid x 4 weeks; up-titrated to 125mg bid x 20 weeks
  Interventions: Drug: Bosentan

INTERVENTIONS:
Drug: Bosentan — Bosentan 62.5mg bid x 4 weeks; up-titrated to 125mg bid x 20 weeks

SUMMARY:
Systemic sclerosis (SSc) is a connective tissue disease characterized by excessive collagen deposition, autoimmunity and by vascular hyper-reactivity and obliterative microvascular phenomena that involves multiple organs. Scleroderma Renal Crisis (SRC) occurs in 5% of patients and mainly with diffuse cutaneous SSc. The routine use of angiotensin-converting enzyme inhibitors (ACEI) has been reported to dramatically improve outcome, with a fall of the 12-month mortality from 76% to less than 15% in the United-States. Despite prognostic improvement, SRC remains a severe manifestation of SSc and functional outcome and survival remains poor. Bosentan is a specific, orally active, dual endothelin receptor antagonist that has recently been approved for the treatment of primary pulmonary arterial hypertension and for the prevention of ischemic digital ulcers. Bosentan could have therapeutic benefits on others vascular injuries and particularly in SRC.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a connective tissue disease characterized by excessive collagen deposition, autoimmunity and by vascular hyper-reactivity and obliterative microvascular phenomena that involves multiple organs. Scleroderma Renal Crisis (SRC) occurs in 5% of patients and mainly with diffuse cutaneous SSc. The routine use of angiotensin-converting enzyme inhibitors (ACEI) has been reported to dramatically improve outcome, with a fall of the 12-month mortality from 76% to less than 15% in the United-States. Despite prognostic improvement, SRC remains a severe manifestation of SSc and functional outcome and survival remains poor. Bosentan is a specific, orally active, dual endothelin receptor antagonist that has recently been approved for the treatment of primary pulmonary arterial hypertension and for the prevention of ischemic digital ulcers. Bosentan could have therapeutic benefits on others vascular injuries and particularly in SRC.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 years
* Patients had to fulfil ACR and/or LEROY et MEDSGER criteria for systemic sclerosis
* Patients had to fulfil criteria for renal systemic sclerosis
* Written informed consent obtained

Exclusion Criteria:

* Scleroderma renal crisis occuring before the age of eighteen
* Patients who are receiving bosentan within one month of inclusion for pulmonary arterial hypertension or digital ulcers prevention
* Other treatment by selective or nonselective antagonist endothelin receptor
* Left ventricle systolic dysfunction (EF < 40 %)
* Patients with systolic blood pressure < 85mm Hg
* Progressive cancer or considered cured for less than 5 years
* Patients with a known hypersensitivity to bosentan or any of the excipients
* Patients with HIV, HCV, HBV infection
* Patients with Liver disease Child-Pugh B and C
* Patients who are pregnant or breast-feeding
* Women of child-bearing age who are sexually active without practising reliable methods of contraception
* Patients who do not give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-12; Primary Completion 2015-10 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
To explore the efficacy of bosentan (Tracleer) in patients with scleroderma renal crisis on renal function | 6 and 12 months

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of bosentan in patients with scleroderma renal crisis over 6 months of treatment | 6 months
1 year overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Alice BEREZNE, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pôle de médecine interne Centre de référence Maladies rares Groupe I Maladies systémiques et maladies auto-immunes rares en particulier Vascularites nécrosantes et les sclérodermies - Hôpital Cochin, Paris, France